CLINICAL TRIAL: NCT01523626
Title: Randomized Study of Early Assessment by CT Scanning in Trauma Patients
Brief Title: A Multicenter, Randomized Study of Early Assessment by CT Scanning in Severely Injured Trauma Patients
Acronym: REACT-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: University Medical Center Nijmegen (Other); Erasmus Medical Center (Other); University Medical Center Groningen (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, J.C. Goslings, Clinical Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1711020323; NTR2607 (Registry Identifier: The Netherlands National Trial Register)
Record Dates: First submitted 2012-01-20; First posted 2012-02-01 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Multiple Trauma/Injuries
Keywords: Trauma; Injur*; Emergen*; Computed Tomography; Total body; TBCT; Whole body; WBCT; Full body; Pan CT
MeSH Terms: conditions — Multiple Trauma; Wounds and Injuries | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional imaging (Other): The control group will be evaluated with X-rays, ultrasonography and selective CT scanning.
  Interventions: Other: Conventional imaging and selective CT scanning.
- Immediate total body CT (Other): The intervention group will receive a 'total body' CT scan from head to pelvis. Conventional radiography and FAST will be completely omitted.
  Interventions: Other: Total body Computed Tomography.

INTERVENTIONS:
Other: Total body Computed Tomography. — The CT protocol for the intervention group consists of a two-step whole-body acquisition (from vertex to pubic symphysis) starting with Head and Neck Non Enhanced CT (NECT) with arms alongside the body.
  The preferred technique for the second complementary scan is a split-bolus intravenous contrast directly after repositioning of the arms alongside the head, and this second scan covers thorax, abdomen and pelvis. Participating centers however are free to choose their own technique as long as intravenous contrast is given for the chest and abdominal part of the TBCT.
  Other Names: Whole body CT; Pan CT; Full body CT; TBCT; WBCT
  Arms: Immediate total body CT
Other: Conventional imaging and selective CT scanning. — The control group will be evaluated according to a conventional trauma protocol with X-rays (of the chest and pelvis), ultrasonography (Focused Assessment with Sonography for Trauma (FAST)) and selective CT scanning.
  Indications for the selective CT scanning are pre-defined and based on the combined local protocols of the participating centers.
  Other Names: X-rays; FAST; Conventional radiography; Computed Tomography; CT
  Arms: Conventional imaging

SUMMARY:
Computed tomography (CT) scanning has become essential in the early diagnostic phase of trauma care because of its high diagnostic accuracy. The introduction of multi-slice CT scanners and infrastructural improvements made 'total body' CT scanning (TBCT) technically feasible and its usage is currently becoming common practice in several trauma centers.

However, literature provides limited evidence whether immediate 'total body' CT scanning leads to better clinical outcome then conventional radiographic imaging supplemented with selective CT scanning in trauma patients. The aim of the REACT-2 trial is to determine the value of immediate TBCT scanning in trauma patients.

The investigators hypothesize that immediate 'total body' CT scanning during the primary survey of severely injured trauma patients has positive effects on patient outcome compared with standard conventional ATLS based radiological imaging supplemented with selective CT scanning.

DETAILED DESCRIPTION:
Injuries are the cause of 5.8 million deaths annually which accounts for almost 10% of global mortality. Among adults aged 15-59 years the proportion of injuries as cause of death is even higher, ranging from 22% to 29% [1].

Specialized trauma centers all over the world provide initial trauma care and diagnostic work-up of trauma patients. This work-up is standardized and frequently based on the Advanced Trauma Life Support (ATLS) guidelines which include a fast and priority-based physical examination as well as screening radiographs supplemented with selective Computed Tomography scanning (CT). ATLS guidelines advise to routinely perform X-rays of thorax and pelvis and Focused Assessment with Sonography for Trauma (FAST) in trauma patients. Whether or not to perform CT scanning following conventional imaging is defined less clearly in the ATLS guidelines and depends upon national guidelines and local protocols.

In recent years CT scanning has become faster, more detailed and more available in the acute trauma care setting. CT shows high accuracy for a wide range of injuries which is reflected by a low missed diagnosis rate. Hence, the conventional radiological work-up according to the ATLS may not be the optimal choice of primary diagnostics anymore. Furthermore, severely injured patients frequently require secondary CT scanning of many parts of the body after conventional imaging. Modern multidetector CT scanners (MDCT) can perform imaging of the head, cervical spine, chest, abdomen and pelvis in a single examination ('total body' CT scanning). The past few years this 'total body' imaging concept gained popularity as a possible alternative to the conventional imaging strategy. With the use of immediate 'total body' CT (TBCT) scanning in trauma patients, rapid and detailed information of organ and tissue injury becomes available and a well-founded plan for further therapy can be made.

In the past, CT scanners were located in the radiology department, frequently even on another floor than the emergency department (ED) were the trauma patient is admitted. The past assumption that TBCT in severely injured trauma patients is too time consuming may no longer be held, since an increasing number of trauma centers have a CT scanner available at the ED or even in the trauma room itself. Several studies evaluated time intervals associated with TBCT usage in severely injured patients. Although these studies are incomparable with respect to design, CT scanners used, diagnostic work-up protocols and trauma populations, the main conclusion is clear. TBCT scanning in trauma patients is not as time consuming as was once expected and may even be time saving compared to conventional imaging protocols supplemented with selective CT.

More and more trauma centers encourage and are implementing immediate TBCT scanning in the diagnostic phase of primary trauma care. Since the burden of TBCT in terms of costs and radiation dose is at least controversial, the advantage of performing immediate TBCT should be proven in high quality studies resulting in high level evidence in order to make its implementation justifiable.

In order to assess the value of immediate TBCT scanning in severely injured trauma patients, the Academic Medical Center (AMC) in Amsterdam, the Netherlands, has initiated an international multicenter randomized clinical trial. Severely injured patients, who are thought to benefit the most from a 'total body' imaging concept, will be included.

ELIGIBILITY:
Inclusion Criteria:

Trauma patient with presence of one of the following criteria:

At least one of the following parameters at hospital arrival:

1. Respiratory rate ≥30/min or ≤10/min
2. Pulse ≥120/min;
3. Systolic blood pressure ≤100 mmHg
4. Estimated external blood loss ≥500 ml
5. Glasgow Coma Score ≤13
6. Abnormal pupillary light reflex.

Or clinical suspicion of one of the following diagnoses:

1. Fractures from at least two long bones
2. Multiple rib fractures, flail chest or open chest
3. Severe abdominal injury
4. Pelvic fracture
5. Unstable vertebral fractures or signs of spinal cord injury.

Or one of the following injury mechanisms:

1. Fall from height (≥ 10 feet)
2. Ejection from the vehicle
3. Death occupant in same vehicle
4. Severely injured patient in same vehicle
5. Wedged or trapped chest / abdomen.

Exclusion Criteria:

1. Age <18 years (if known)
2. Known pregnancy
3. Patients referred from other hospitals
4. Clearly low-energy trauma with blunt injury mechanism
5. Penetrating injury in 1 body region (except gun shot wounds) as the clearly isolated injury
6. Any patient who is judged to be too unstable to undergo a CT scan and requires (cardiopulmonary) resuscitation or immediate operation because death is imminent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1083 (Actual)
Dates: Start 2011-04; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality. | From date of randomization until the date of death from any cause, while being an inpatient, assessed up to 1 year.
  Mortality during hospital admission.

SECONDARY OUTCOMES:
Overall mortality | 24-hour, 30-day and 1-year mortality.
  Mortality in general during specific time frames.
Several clinical relevant time intervals. | From date and time of randomization to date and time of immediate intervention or ICU arrival, with an expected duration of 1-3 hours.
  * time of arrival;
  * time to CT;
  * scanning time;
  * time to diagnosis;
  * time in the trauma room;
  * time to intervention.
Radiation exposure | Until six months posttrauma.
  Radiation dose in miliSievert.
Quality of life | Six and twelve months posttrauma.
  As recorded by completing the EuroQol-6D.
Morbidity | Up to six months posttrauma.
  * complications and total number of (re-)interventions and re-admissions;
  * transfusion requirements;
  * length of ICU stay;
  * number of ventilation days.
General health | Six and twelve months posttrauma.
  As recorded by completing the HUI-3.
Cost-effectiveness analyses. | Until six months posttrauma.
  Cost-effectiveness analyses will be performed with the costs per patient alive and costs per patient alive without serious morbidity as outcome measures.
  Additionally, a cost-utility analysis will be done with the cost per QALY as outcome measure. Incremental cost-effectiveness ratios will be calculated, expressing the extra costs per (i) extra patients alive, (ii) extra patients alive and without serious morbidity, and (iii) additional QALY.

CONTACTS AND LOCATIONS:
Overall Officials: J Carel Goslings, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (5):
- Netherlands (4):
  - Academic Medical Center (AMC), Amsterdam
  - University Medical Center Groningen, Groningen
  - University Medical Centre Nijmegen, Nijmegen
  - Erasmus Medical Center, Rotterdam
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Background] Sethi D, Racioppi F, Baumgarten I, Bertollini R. Reducing inequalities from injuries in Europe. Lancet. 2006 Dec 23;368(9554):2243-50. doi: 10.1016/S0140-6736(06)68895-8. PMID 17189036
- [Background] World Health Organization. The global burden of disease: 2004 update. [http://www.who.int/healthinfo/global_burden_disease/2004_report_update/en/index.html]
- [Background] American College of Surgeons Committee on Trauma.: ATLS advanced trauma life support program for doctors. Student Course Manual., 8th. edn. Chigago, IL: 2008.
- [Background] Albrecht T, von Schlippenbach J, Stahel PF, Ertel W, Wolf KJ. [The role of whole body spiral CT in the primary work-up of polytrauma patients--comparison with conventional radiography and abdominal sonography]. Rofo. 2004 Aug;176(8):1142-50. doi: 10.1055/s-2004-813259. German. PMID 15346611
- [Background] Brenner DJ, Elliston CD. Estimated radiation risks potentially associated with full-body CT screening. Radiology. 2004 Sep;232(3):735-8. doi: 10.1148/radiol.2323031095. Epub 2004 Jul 23. PMID 15273333
- [Background] Deunk J, Brink M, Dekker HM, Kool DR, van Kuijk C, Blickman JG, van Vugt AB, Edwards MJ. Routine versus selective computed tomography of the abdomen, pelvis, and lumbar spine in blunt trauma: a prospective evaluation. J Trauma. 2009 Apr;66(4):1108-17. doi: 10.1097/TA.0b013e31817e55c3. PMID 19359922
- [Background] Fanucci E, Fiaschetti V, Rotili A, Floris R, Simonetti G. Whole body 16-row multislice CT in emergency room: effects of different protocols on scanning time, image quality and radiation exposure. Emerg Radiol. 2007 Feb;13(5):251-7. doi: 10.1007/s10140-006-0554-0. Epub 2006 Dec 20. PMID 17180674
- [Background] Gralla J, Spycher F, Pignolet C, Ozdoba C, Vock P, Hoppe H. Evaluation of a 16-MDCT scanner in an emergency department: initial clinical experience and workflow analysis. AJR Am J Roentgenol. 2005 Jul;185(1):232-8. doi: 10.2214/ajr.185.1.01850232. PMID 15972429
- [Background] Hilbert P, zur Nieden K, Hofmann GO, Hoeller I, Koch R, Stuttmann R. New aspects in the emergency room management of critically injured patients: a multi-slice CT-oriented care algorithm. Injury. 2007 May;38(5):552-8. doi: 10.1016/j.injury.2006.12.023. PMID 17472791
- [Background] Huber-Wagner S, Lefering R, Qvick LM, Korner M, Kay MV, Pfeifer KJ, Reiser M, Mutschler W, Kanz KG; Working Group on Polytrauma of the German Trauma Society. Effect of whole-body CT during trauma resuscitation on survival: a retrospective, multicentre study. Lancet. 2009 Apr 25;373(9673):1455-61. doi: 10.1016/S0140-6736(09)60232-4. Epub 2009 Mar 25. PMID 19321199
- [Background] Kalender WA, Seissler W, Klotz E, Vock P. Spiral volumetric CT with single-breath-hold technique, continuous transport, and continuous scanner rotation. Radiology. 1990 Jul;176(1):181-3. doi: 10.1148/radiology.176.1.2353088.
- [Background] Kanz KG, Korner M, Linsenmaier U, Kay MV, Huber-Wagner SM, Kreimeier U, Pfeifer KJ, Reiser M, Mutschler W. [Priority-oriented shock trauma room management with the integration of multiple-view spiral computed tomography]. Unfallchirurg. 2004 Oct;107(10):937-44. doi: 10.1007/s00113-004-0845-4. German. PMID 15452654
- [Background] Kanz KG, Paul AO, Lefering R, Kay MV, Kreimeier U, Linsenmaier U, Mutschler W, Huber-Wagner S; Trauma Registry of the German Trauma Society. Trauma management incorporating focused assessment with computed tomography in trauma (FACTT) - potential effect on survival. J Trauma Manag Outcomes. 2010 May 10;4:4. doi: 10.1186/1752-2897-4-4. PMID 20459713
- [Background] Kim PK, Gracias VH, Maidment AD, O'Shea M, Reilly PM, Schwab CW. Cumulative radiation dose caused by radiologic studies in critically ill trauma patients. J Trauma. 2004 Sep;57(3):510-4. doi: 10.1097/01.ta.0000141028.97753.67. PMID 15454795
- [Background] Leidner B, Adiels M, Aspelin P, Gullstrand P, Wallen S. Standardized CT examination of the multitraumatized patient. Eur Radiol. 1998;8(9):1630-8. doi: 10.1007/s003300050601. PMID 9866776
- [Background] Linsenmaier U, Krotz M, Hauser H, Rock C, Rieger J, Bohndorf K, Pfeifer KJ, Reiser M. Whole-body computed tomography in polytrauma: techniques and management. Eur Radiol. 2002 Jul;12(7):1728-40. doi: 10.1007/s00330-001-1225-x. Epub 2001 Dec 13. PMID 12111064
- [Background] Low R, Duber C, Schweden F, Lehmann L, Blum J, Thelen M. [Whole body spiral CT in primary diagnosis of patients with multiple trauma in emergency situations]. Rofo. 1997 May;166(5):382-8. doi: 10.1055/s-2007-1015446. German. PMID 9198509
- [Background] Maurer MH, Knopke S, Schroder RJ. [Added diagnostic benefit of 16-row whole-body spiral CT in patients with multiple trauma differentiated by region and injury severity according to the ATLS concept]. Rofo. 2008 Dec;180(12):1117-23. doi: 10.1055/s-2008-1027851. Epub 2008 Nov 28. German. PMID 19235701
- [Background] Nguyen D, Platon A, Shanmuganathan K, Mirvis SE, Becker CD, Poletti PA. Evaluation of a single-pass continuous whole-body 16-MDCT protocol for patients with polytrauma. AJR Am J Roentgenol. 2009 Jan;192(1):3-10. doi: 10.2214/AJR.07.3702. PMID 19098172
- [Background] Philipp MO, Kubin K, Hormann M, Metz VM. Radiological emergency room management with emphasis on multidetector-row CT. Eur J Radiol. 2003 Oct;48(1):2-4. doi: 10.1016/s0720-048x(03)00206-7. PMID 14511855
- [Background] Prokop A, Hotte H, Kruger K, Rehm KE, Isenberg J, Schiffer G. [Multislice CT in diagnostic work-up of polytrauma]. Unfallchirurg. 2006 Jul;109(7):545-50. doi: 10.1007/s00113-006-1086-5. German. PMID 16636783
- [Background] Ptak T, Rhea JT, Novelline RA. Radiation dose is reduced with a single-pass whole-body multi-detector row CT trauma protocol compared with a conventional segmented method: initial experience. Radiology. 2003 Dec;229(3):902-5. doi: 10.1148/radiol.2293021651. PMID 14657320
- [Background] Rieger M, Sparr H, Esterhammer R, Fink C, Bale R, Czermak B, Jaschke W. [Modern CT diagnosis of acute thoracic and abdominal trauma]. Anaesthesist. 2002 Oct;51(10):835-42. doi: 10.1007/s00101-002-0369-7. German. PMID 12395175
- [Background] Rieger M, Czermak B, El Attal R, Sumann G, Jaschke W, Freund M. Initial clinical experience with a 64-MDCT whole-body scanner in an emergency department: better time management and diagnostic quality? J Trauma. 2009 Mar;66(3):648-57. doi: 10.1097/TA.0b013e31816275f3. PMID 19276733
- [Background] Ruchholtz S, Waydhas C, Schroeder T, Piepenbrink K, Kuhl H, Nast-Kolb D. [The value of computed tomography in the early treatment of seriously injured patients]. Chirurg. 2002 Oct;73(10):1005-12. doi: 10.1007/s00104-002-0429-1. German. PMID 12395159
- [Background] Salim A, Sangthong B, Martin M, Brown C, Plurad D, Demetriades D. Whole body imaging in blunt multisystem trauma patients without obvious signs of injury: results of a prospective study. Arch Surg. 2006 May;141(5):468-73; discussion 473-5. doi: 10.1001/archsurg.141.5.468. PMID 16702518
- [Background] Saltzherr TP, Goslings JC; multidisciplinary REACT 2 study group. Effect on survival of whole-body CT during trauma resuscitation. Lancet. 2009 Jul 18;374(9685):198; author reply 198-9. doi: 10.1016/S0140-6736(09)61324-6. No abstract available. PMID 19616711
- [Background] Sampson MA, Colquhoun KB, Hennessy NL. Computed tomography whole body imaging in multi-trauma: 7 years experience. Clin Radiol. 2006 Apr;61(4):365-9. doi: 10.1016/j.crad.2005.12.009. PMID 16546467
- [Background] Smith CM, Woolrich-Burt L, Wellings R, Costa ML. Major trauma CT scanning: the experience of a regional trauma centre in the UK. Emerg Med J. 2011 May;28(5):378-82. doi: 10.1136/emj.2009.076414. Epub 2010 Jun 1. PMID 20515906
- [Background] Tien HC, Tremblay LN, Rizoli SB, Gelberg J, Spencer F, Caldwell C, Brenneman FD. Radiation exposure from diagnostic imaging in severely injured trauma patients. J Trauma. 2007 Jan;62(1):151-6. doi: 10.1097/TA.0b013e31802d9700. PMID 17215747
- [Background] Weninger P, Mauritz W, Fridrich P, Spitaler R, Figl M, Kern B, Hertz H. Emergency room management of patients with blunt major trauma: evaluation of the multislice computed tomography protocol exemplified by an urban trauma center. J Trauma. 2007 Mar;62(3):584-91. doi: 10.1097/01.ta.0000221797.46249.ee. PMID 17414332
- [Background] Wurmb T, Fruhwald P, Brederlau J, Steinhubel B, Frommer M, Kuhnigk H, Kredel M, Knupffer J, Hopfner W, Maroske J, Moll R, Wagner R, Thiede A, Schindler G, Roewer N. [The Wurzburg polytrauma algorithm. Concept and first results of a sliding-gantry-based computer tomography diagnostic system]. Anaesthesist. 2005 Aug;54(8):763-8; 770-2. doi: 10.1007/s00101-005-0850-1. German. PMID 15959743
- [Background] Wurmb T, Balling H, Fruhwald P, Keil T, Kredel M, Meffert R, Roewer N, Brederlau J. [Polytrauma management in a period of change: time analysis of new strategies for emergency room treatment]. Unfallchirurg. 2009 Apr;112(4):390-9. doi: 10.1007/s00113-008-1528-3. German. PMID 19159120
- [Background] Wurmb TE, Fruhwald P, Hopfner W, Keil T, Kredel M, Brederlau J, Roewer N, Kuhnigk H. Whole-body multislice computed tomography as the first line diagnostic tool in patients with multiple injuries: the focus on time. J Trauma. 2009 Mar;66(3):658-65. doi: 10.1097/TA.0b013e31817de3f4. PMID 19276734
- [Background] Wurmb TE, Quaisser C, Balling H, Kredel M, Muellenbach R, Kenn W, Roewer N, Brederlau J. Whole-body multislice computed tomography (MSCT) improves trauma care in patients requiring surgery after multiple trauma. Emerg Med J. 2011 Apr;28(4):300-4. doi: 10.1136/emj.2009.082164. Epub 2010 Jul 20. PMID 20659885
- [Derived] Treskes K, Saltzherr TP, Edwards MJR, Beuker BJA, Den Hartog D, Hohmann J, Luitse JS, Beenen LFM, Hollmann MW, Dijkgraaf MGW, Goslings JC; REACT-2 study group. Emergency Bleeding Control Interventions After Immediate Total-Body CT Scans in Trauma Patients. World J Surg. 2019 Feb;43(2):490-496. doi: 10.1007/s00268-018-4818-0. PMID 30327841
- [Derived] Sierink JC, Treskes K, Edwards MJ, Beuker BJ, den Hartog D, Hohmann J, Dijkgraaf MG, Luitse JS, Beenen LF, Hollmann MW, Goslings JC; REACT-2 study group. Immediate total-body CT scanning versus conventional imaging and selective CT scanning in patients with severe trauma (REACT-2): a randomised controlled trial. Lancet. 2016 Aug 13;388(10045):673-83. doi: 10.1016/S0140-6736(16)30932-1. Epub 2016 Jun 28. PMID 27371185
- [Derived] Hajibandeh S, Hajibandeh S. Systematic review: effect of whole-body computed tomography on mortality in trauma patients. J Inj Violence Res. 2015 Jul;7(2):64-74. doi: 10.5249/jivr.v7i2.613. PMID 26104319
- [Derived] Sierink JC, Saltzherr TP, Beenen LF, Luitse JS, Hollmann MW, Reitsma JB, Edwards MJ, Hohmann J, Beuker BJ, Patka P, Suliburk JW, Dijkgraaf MG, Goslings JC; REACT-2 study group. A multicenter, randomized controlled trial of immediate total-body CT scanning in trauma patients (REACT-2). BMC Emerg Med. 2012 Mar 30;12:4. doi: 10.1186/1471-227X-12-4. PMID 22458247